CLINICAL TRIAL: NCT06098716
Title: All in the Family: Promoting Family Function Through Physical Activity
Acronym: SSHRC-Family
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 435-2023-0493
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Physical Activity; Family Functioning
Keywords: Parenting Practices; Exercise; Family Functioning; Identity; Self-Regulation;; Parental Support
MeSH Terms: conditions — Motor Activity; Self-Control | interventions — Professional Autonomy; Educational Status

STUDY DESIGN:
Intervention Model Description: 3 arm parallel design single blinded randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Education (Active Comparator): The Education condition package will consist of Canada's PA guidelines, information about the benefits of child and adult PA, healthy living and a breakdown of ways for the parent to help their child achieve this PA.
  Interventions: Behavioral: Education
- Self Regulation (Experimental): The SR condition will receive all of the same education material as the education condition in addition to skill training content (how to plan for family PA) based on our prior family trials. Families will be instructed to plan for "when," "where," "how," and "what" PA will be performed, and to create back-up plans commensurate with the creation of action and coping planning.
  Interventions: Behavioral: Self Regulation; Behavioral: Education
- PA Support & Family Social Identity (Experimental): The ID condition receives the same education and self-regulation content as the other groups, but with additional activities designed to strengthen (i) parents' PA-support identity and (ii) the family's shared PA social identity. Session 1 involves only the parent(s) and focuses on parental support identity. The content is based on the behaviour change principles of self-identity theory that should lead to increases in self-identity. This session's activities include: 1) bringing awareness to the concept of identity and being a role model, 2) an activity on finding the meaning and value of parental support of child PA, 3) an activity on setting prioritization rules around parental support for child PA in comparison to other parenting responsibilities and values (brainstormed), 4) developing an affirmation for parental support self-talk, and 5) planning ways to visually demonstrate the parental support identity for self-categorization (e.g., on social media, pictures in frames).
  Interventions: Behavioral: Self Regulation; Behavioral: PA Support & Family Social Identity; Behavioral: Education

INTERVENTIONS:
Behavioral: Self Regulation — How to plan for Family PA
  Arms: PA Support & Family Social Identity; Self Regulation
Behavioral: PA Support & Family Social Identity — Exercises that strengthen parents' PA-support identity and a shared active-family identity through values reflection, role-modelling, visualization, and visible "active family" cues.
  Arms: PA Support & Family Social Identity
Behavioral: Education — Information about healthy living (e.g., PA, sleep hygiene and healthy eating)

SUMMARY:
The goal of this trial is to find out whether adding identity-building and self-regulation training to basic healthy-living education helps families with inactive children (ages 6-12) become more cohesive and physically active. The main question it aims to answer is:

Does the identity + self-regulation + education program improve family cohesion more than (a) self-regulation + education or (b) education alone?

Researchers will compare three groups-identity+self-regulation+education (ID), self-regulation+education (SR), and education-only (ED)-to see which produces the greatest improvements.

Participants will:

1. attend three online workshops at baseline plus two booster sessions at 6-week and 3-month with a project coordinator;
2. complete online questionnaires at baseline, 6-week, 3-month, and 6-month;
3. take part in an exit interview at 6 months.

DETAILED DESCRIPTION:
The primary objective of this study is to test the efficacy of three family physical activity (PA) interventions on a key family functioning outcome-family cohesion-through increased PA in children and parent-child co-PA. Our study tests three intervention conditions: 1) identity (ID; promotion of a PA parenting identities + self-regulation skills + education), 2) self-regulation (SR; promotion of PA parenting self-regulation skills + education) and 3) education (ED; an education about PA control condition). It is hypothesised that (H1): The ID condition will show significantly larger changes in family cohesion compared to the two other conditions after six-months (primary end-point) and (H2): The SR condition will show significantly larger changes in family cohesion compared to the ED control condition after six-months.

There are three secondary objectives for this study. First, this study aims to assess the impact of the three interventions on the remaining family-functioning dimensions-flexibility and organisation-and on behavioural outcomes (child MVPA and parent-child co-PA) at the 6-month end-point. The ID condition is hypothesized to lead to significantly greater increases in family flexibility, family organization, child MVPA and parent-child co-PA compared to the SR and ED conditions after six months (H3), with the SR condition also expected to outperform the ED condition in these PA outcomes (H4).

Second, this study will also investigate whether group differences in child and parent PA and family functioning outcomes can be explained through a mediation model based on the Multi-Process Action Control (M-PAC) framework. It is hypothesized that changes in child MVPA and parent-child co-PA will mediate the relationship between the intervention groups and family functioning outcomes. These changes in PA behaviors are expected to be predicted by alterations in family social identity and parental PA support identity, which will, in turn, be influenced by parental attitudes, perceptions of control (reflective processes), and behavioral self-regulation (regulatory processes) regarding child PA (H5).

Third, the present study will explore the potential moderating effects of seasonal variation, child sex, dual/single-parent status, parent sex and gender, child age, intervention adherence, and the type and format of PA on the primary outcomes across the three intervention conditions. While no specific hypotheses are pre-set for these factors, it is anticipated that participation in PA may decrease during winter due to weather conditions, and single-parent families might face more barriers to parent-child co-PA, leading to lower participation levels. Additionally, the composition and frequency patterns of child MVPA may influence family functioning outcomes differently across the intervention conditions.

ELIGIBILITY:
Inclusion Criteria:

Participants will be at least one parent with at least one child between the ages of 6 and 12 years.

Families (parents and/or guardians and children) residing in Canada. Children that participate in <60 minutes/day of moderate to vigorous physical activity (MVPA).

Exclusion Criteria:

If child is meeting the current physical activity guidelines >=60 minutes a day of moderate to vigorous physical activity per day.

If the participant does not pass the Physical Activity Readiness Questionnaire (PARQ) If children's age falls outside the 6-12 year range

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Family cohesion | Baseline, 6 weeks, 3 months, and 6 months
  Family cohension will be assessed using FAD & FACES IV subscale = 1 = Strongly Disagree; 2 = Generally Disagree; 3 = Undecided; 4 = Generally Agree; 5 = Strongly Agree

SECONDARY OUTCOMES:
Family functioning outcomes (i.e., family organisation and flexibility) | Baseline, 6 weeks, 3 months, and 6 months
  Family organisation and flexibility will be assessed using FAD & FACES IV subscale = 1 = Strongly Disagree; 2 = Generally Disagree; 3 = Undecided; 4 = Generally Agree; 5 = Strongly Agree
Children's moderate to vigorous physical activity (MVPA) | Baseline, 6 weeks, 3 months, and 6 months
  Children's physical activity will be quantified by Self Report using Physical Activity Questionnaire for Children (PAQ-C)
Parent-child intergenerational activity measured via parent self-report | Baseline, 6 weeks, 3 months, and 6 months
  For parent-child co-PA, the Godin Leisure-Time Exercise Questionnaire will be used.
Parental support and M-PAC Constructs | Baseline, 6 weeks, 3 months, and 6 months
  Parental support for child PA: 6-item activity-related parenting practices scale Parental support identity: 3-item version of the Exercise Identity Scale Family PA identity: 4-item scale from Doosje, Ellemers 's ingroup identification measure Parental support habits: 4-item version of the Self-Reported Habit Strength Index Behavioral regulation of parental support: 11-item Physical Activity Regulation Scale Perceived capability and perceived opportunity: 7-item perceived control measure Attitude: 6-item affective and instrumental attitude scale Parental intention: 2-item decisional intention and intention strength scale

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee ASY, Blanchard CM, Beauchamp MR, Carson V, Madigan S, Strachan S, Vanderloo LM, Streight E, Courtnall S, Rhodes RE. Promoting family functioning through physical activity: a randomized trial to evaluate the "All in the Family" program. Trials. 2025 Aug 12;26(1):287. doi: 10.1186/s13063-025-08977-6. PMID 40796896